CLINICAL TRIAL: NCT01359163
Title: An Open Label, Randomized, Single Dose, Crossover Pivotal Bioequivalence Study Of Commercial Femulen Tablets Versus Reformulated Femulen Tablets In Healthy Female Subjects
Brief Title: A Study To Determine Bioequivalence Between The Commercial Femulen Tablets And A Reformulation Of Femulen Tablets In Healthy Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B1361002
Record Dates: First submitted 2011-05-20; First posted 2011-05-24 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-04

CONDITIONS: Therapeutic Equivalency
Keywords: bioequivalence study; marketed vs reformulation tablets; Femulen
MeSH Terms: interventions — Ethynodiol Diacetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Femulen commercial tablets (Active Comparator)
  Interventions: Drug: etynodiol diacetate
- Femulen reformulated tablets (Experimental)
  Interventions: Drug: etynodiol diacetate

INTERVENTIONS:
Drug: etynodiol diacetate — tablet, 0.5 mg, single dose
  Arms: Femulen commercial tablets
Drug: etynodiol diacetate — tablet, 0.5 mg, single dose
  Arms: Femulen reformulated tablets

SUMMARY:
A pivotal study to determine bioequivalence between a the current marketed formulation of Femulen tablets and reformulated Femulen tablets in healthy female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >45 kg (99 lbs).
* Healthy female subjects between the ages of 21 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).

Ages: 21 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Area under the curve to last time point observed (AUCt) | 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48
Highest concentration (Cmax) | 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48

SECONDARY OUTCOMES:
Area under the curve to infinity (AUCinf) | 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48
Area under the curve percent to infinity (AUC%inf) | 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48
Half-life (T1/2) | 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48
Time at maximum concentration (Tmax) | 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1361002&StudyName=A%20Study%20To%20Determine%20Bioequivalence%20Between%20The%20Commercial%20Femulen%20Tablets%20And%20A%20Reformulation%20Of%20Femulen%20Tablets%20In%20Healthy%20Female%20Subj